CLINICAL TRIAL: NCT00245518
Title: Effect of Isoflavones on Cognition, Quality of Life and Hot Flashes in Men With Prostate Cancer Undergoing Androgen Deprivation Therapy
Brief Title: Effect of Soy on Cognition and Hot Flashes in Men With Prostate Cancer Undergoing Testosterone Suppression Therapy
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Johns Hopkins University (Other)
Collaborators: Physicians Laboratories (Unknown); National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Double | Purpose: Treatment
Other Study IDs: 04-08-09-04
Record Dates: First submitted 2005-10-26; First posted 2005-10-28 (Estimated); Results first posted 2017-10-13 (Actual); Last update posted 2017-10-13 (Actual); Status verified 2017-09

CONDITIONS: Hot Flashes
Keywords: prostate cancer; soy; androgen deprivation; quality of life; isoflavones
MeSH Terms: conditions — Hot Flashes; Prostatic Neoplasms | interventions — Isoflavones

STUDY DESIGN:
Who Masked: Participant, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Isoflavone (Experimental): Isoflavone
  Interventions: Drug: Isoflavone
- Placebo (Placebo Comparator)
  Interventions: Drug: Placebos

INTERVENTIONS:
Drug: Isoflavone
  Arms: Isoflavone
Drug: Placebos
  Arms: Placebo

SUMMARY:
This study will look at the effects of a soy supplement called Revival on memory, quality of life, and hot flashes in men with prostate cancer who are being treated with testosterone suppression therapy. Hypothesis: Treating men who have prostate CA with daily Revival will result in at least a 50% reduction in hot flashes compared to placebo.

DETAILED DESCRIPTION:
This research study will look at the effects of a soy supplement called Revival on memory, quality of life, and hot flashes in men with prostate cancer who are undergoing (ADT) androgen deprivation therapy. Participants will be given either placebo or Revival. Participants will be asked to take their supplement once/day for 14 weeks.Blood will be drawn to check on liver, kidney, thyroid, cholesterol,and prostate health. Urine will be collected to check on bone markers. Patients will be asked to complete questionnaires to test memory, attention span, and vocabulary.Possible benefits may include increase in memory, decrease in hot flashes, and a general increase in quality of life.

ELIGIBILITY:
Inclusion Criteria:

* men > or =21 with prostate CA and hypogonadism for at least 3 months

Exclusion Criteria:

* on growth promoting agents
* on appetite stimulating agents
* on Prednisone and others

Min Age: 21 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2005-06; Primary Completion 2008-09 (Actual); Study Completion 2008-09 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Shehzad Basaria, M.D., Principal Investigator — Johns Hopkins University
Locations (1):
- Johns Hopkins University Clinical Trials Unit, Baltimore, Maryland, United States

RESULTS

PARTICIPANT FLOW:
Pre-assignment Details: 39 participants were enrolled in this study. 3 were not randomized due to failed screening on laboratory assessment, 2 because they withdrew due to personal reasons, and 1 because of dislike of the taste of the compound.
Groups:
- Placebo: Placebos
Period: Overall Study
Arm/Group | Isoflavone | Placebo
Started | 17 | 16
Completed | 17 | 16
Not Completed | 0 | 0

BASELINE CHARACTERISTICS:
Population: Baseline characteristics were only recorded for the 33 participants who completed the study.
Groups:
- Total: Total of all reporting groups
Arm/Group | Isoflavone | Placebo | Total
Number analyzed (Participants) | 17 | 16 | 33
Age, Customized [Count of Participants; unit: Participants]
  >= 21 years | 17 | 16 | 33
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 0 | 0 | 0
  Male | 17 | 16 | 33
Region of Enrollment [Count of Participants; unit: Participants]
  United States | 17 | 16 | 33

OUTCOME MEASURES:

1. Primary Outcome: Cognitive Function as Assessed by the National Adult Reading Test (NART)
Description: the NART estimates intelligence levels of English-speaking patients. It consists of 50 short words with irregular spelling or phonetic appearance which the participant must read and pronounce. The higher the score, the higher number of correct responses. Scores are 0-50.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Groups:
- Placebo: Placebo
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 45.2 (2.12) | 39.6 (3.02)
  6 weeks | 42.43 (2.66) | 41.29 (3.25)
  12 weeks | 43.69 (2.83) | 41.57 (3.21)

2. Primary Outcome: Cognitive Function as Assessed by the Hopkins Verbal Learning Test (HVLT), Total Recall Score
Description: The test consists 12 nouns, four words each from one of three semantic categories (e.g., precious gems, articles of clothing, vegetables, etc.), to be learned over the course of three learning trials. Approximately 20-25 min later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives, 6 semantically related, & 6 semantically unrelated. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score ( -12) ; the retention (%) score (0-100%) is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher score = higher cognition.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 24.67 (1.67) | 21.6 (1.26)
  6 weeks | 24.87 (1.57) | 22.53 (0.96)
  12 weeks | 25.85 (1.56) | 22.47 (1.39)

3. Primary Outcome: Cognitive Function as Assessed by the Hopkins Verbal Learning Test (HVLT), Recognition Discrimination Index
Description: The test consists 12 nouns, four words each from one of three semantic categories (e.g., precious gems, articles of clothing, vegetables, etc.), to be learned over the course of three learning trials. Approximately 20-25 min later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives, 6 semantically related, & 6 semantically unrelated. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score ( -12) ; the retention (%) score (0-100%) is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives. A higher score= higher cognitive function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 22.13 (0.46) | 20.8 (0.87)
  6 weeks | 20.4 (1) | 21.47 (1)
  12 weeks | 22.77 (0.53) | 22.67 (0.67)

4. Primary Outcome: Cognitive Function as Assessed by the Hopkins Verbal Learning Test (HVLT), Percent Retained
Description: The test consists 12 nouns, four words each from one of three semantic categories (e.g., precious gems, articles of clothing, vegetables, etc.), to be learned over the course of three learning trials. Approximately 20-25 min later, a delayed recall trial and a recognition trial are completed. The delayed recall requires free recall of any words remembered. The recognition trial is composed of 24 words, including the 12 target words and 12 false-positives, 6 semantically related, and 6 semantically unrelated. When scoring the HVLT, the three learning trials are combined to calculate a total recall score (0-36); the delayed recall trial creates the delayed recall score ( -12) ; the retention (%) score (0-100%) is calculated by dividing the delayed recall trial by the higher of learning trial 2 or 3; and the recognition discrimination index is comprised by subtracting the total number of false positives from the total number of true positives.A higher score= higher cognitive function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 100.88 (5.98) | 89.82 (5.84)
  6 weeks | 94.31 (2.38) | 94.08 (4.3)
  12 weeks | 94.68 (3.63) | 95.21 (5.5)

5. Primary Outcome: Cognitive Function as Assessed by the F-A-S Test
Description: The F-A-S Test, a subtest of the Neurosensory Center Comprehensive Examination for Aphasia (NCCEA), is a measure of phonemic word fluency, which is a type of verbal fluency. It assesses phonemic fluency by requesting an individual to orally produce as many words as possible that begin with the letters F, A, and S within a prescribed time frame (1 minute)
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: seconds
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
seconds
  Baseline | 58.79 (3.65) | 55.36 (5.08)
  6 weeks | 64.47 (4.51) | 56.93 (4.78)
  12 weeks | 63.31 (4.43) | 57.93 (4.42)

6. Primary Outcome: Cognition as Assessed by the Grooved Pegboard Test (GPT) , Dominant Hand Time (Seconds)
Description: The GPT assesses eye-hand coordination and motor speed and thus requires sensory motor integration and a high level of motor processing. The test apparatus consists of a square metal surface (10.1 cm2) with a 5 × 5 matrix of keyhole shaped holes in various orientations. The task requires the examinee to pick up the keyhole shaped peg (3 mm in diameter) individually from the well just above the 5 × 5 matrix of holes from left to right and top to bottom as quickly as possible using the dominant hand. Because the holes are in various orientations, examinees must manipulate each peg in their hand (usually between the index finger and thumb) so that the peg aligns with the orientation of the hole. A faster time, indicates greater cognitive functioning.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
time in seconds
  Baseline | 101.5 (8.14) | 91.8 (8.7)
  6 weeks | 89.93 (4.32) | 78.73 (3.34)
  12 weeks | 90.75 (6.05) | 83.8 (5.72)

7. Primary Outcome: Cognition as Assessed by the Grooved Pegboard Test (GPT) , Non-dominant Hand Time (Seconds)
Description: The GPT assesses eye-hand coordination and motor speed and thus requires sensory motor integration and a high level of motor processing. The test apparatus consists of a square metal surface (10.1 cm2) with a 5 × 5 matrix of keyhole shaped holes in various orientations. The task requires the examinee to pick up the keyhole shaped peg (3 mm in diameter) individually from the well just above the 5 × 5 matrix of holes from left to right and top to bottom as quickly as possible using the non-dominant hand. Because the holes are in various orientations, examinees must manipulate each peg in their hand (usually between the index finger and thumb) so that the peg aligns with the orientation of the hole.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: time in seconds
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
time in seconds
  Baseline | 115.43 (9.75) | 112.8 (11.25)
  6 weeks | 98.86 (7.76) | 89.2 (3.05)
  12 weeks | 102.73 (7.43) | 88.67 (6.91)

8. Primary Outcome: Cognition as Assessed by the Grooved Pegboard Test (GPT) , Number of Dominant Hand Drops
Description: The GPT assesses eye-hand coordination and motor speed and thus requires sensory motor integration and a high level of motor processing. The test apparatus consists of a square metal surface (10.1 cm2) with a 5 × 5 matrix of keyhole shaped holes in various orientations. The task requires the examinee to pick up the keyhole shaped peg (3 mm in diameter) individually from the well just above the 5 × 5 matrix of holes from left to right and top to bottom as quickly as possible using the dominant hand. Because the holes are in various orientations, examinees must manipulate each peg in their hand (usually between the index finger and thumb) so that the peg aligns with the orientation of the hole.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: number of times peg dropped
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
number of times peg dropped
  Baseline | 0.64 (0.27) | 0.4 (0.19)
  6 weeks | 0.14 (0.1) | 0.33 (0.21)
  12 weeks | 0.09 (0.09) | 0.2 (0.11)

9. Primary Outcome: Cognition as Assessed by the Grooved Pegboard Test (GPT) , Number of Non- Dominant Hand Drops
Description: as for outcome 8
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: number of times peg dropped
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
number of times peg dropped
  Baseline | 0.21 (0.11) | 0.6 (0.4)
  6 weeks | 0.07 (0.07) | 0.4 (0.13)
  12 weeks | 0.45 (0.28) | 0.27 (0.12)

10. Primary Outcome: Cognition as Assessed by the Rex Complex Figure Test (RCFT), Immediate Recall
Description: The test measures recognition memory for the elements of the Rey complex figure, and assesses the respondent's ability to use cues to retrieve information. Scoring of drawings is based on the widely used 36-point scoring system. Each of the 18 scoring units is scored based on accuracy and placement criteria. Items of the figure can earn points:
  1. Correct Image: placed properly (2 points), placed poorly (1 point)
  2. Distorted or Incomplete Image, but recognizable: placed properly (1 point), placed poorly (1/2) point
  3. Absent or not recognizable: 0 points
  Scale ranges 0-36. with 36 being greatest cognitive function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 20.87 (1.15) | 16.03 (2.21)
  6 weeks | 24.33 (1.4) | 22.33 (1.62)
  12 weeks | 25.92 (1.52) | 25.13 (1.91)

11. Primary Outcome: Cognition as Assessed by the Rex Complex Figure Test (RCFT), Delayed Recall
Description: The test measures recognition memory for the elements of the Rey complex figure, and assesses the respondent's ability to use cues to retrieve information after 25-30 minutes. Scoring of drawings is based on the widely used 36-point scoring system. Each of the 18 scoring units is scored based on accuracy and placement criteria. Items of the figure can earn points:
  1. Correct Image: placed properly (2 points), placed poorly (1 point)
  2. Distorted or Incomplete Image, but recognizable: placed properly (1 point), placed poorly (1/2) point
  3. Absent or not recognizable: 0 points
  Scale ranges 0-36, with 36 representing maximum cognition .
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 20.37 (1.44) | 23.07 (1.43)
  6 weeks | 23.07 (1.43) | 20.43 (1.61)
  12 weeks | 24.42 (1.79) | 24.27 (2.04)

12. Primary Outcome: Sexual Function as Assessed by the Watts Sexual Function Questionnaire (WSFQ), Total Score
Description: The WSFQ contains 17 items that assess the domains of sexual desire/libido (6 items), arousal (1 item), orgasm/erectile function (7 items), and satisfaction(3 items). A five-point Likert-type scale ranging from "always" to "never" is used to generate a total score and four domain scores. The possible range of total sexual function scores is 17 to 85. Higher scores indicate better sexual function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 62.92 (3.18) | 62 (3.71)
  6 weeks | 63.21 (2.3) | 63.83 (2.79)
  12 weeks | 59.7 (3.39) | 67 (3.68)

13. Primary Outcome: Sexual Function as Assessed by the Watts Sexual Function Questionnaire (WSFQ), Libido
Description: The domain of sexual desire/libido consists of 6 items. A five-point Likert-type scale ranging from "always" to "never" is used to generate a score, ranging from 6-30. Higher scores indicate increased libido/sexual desire.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 22.21 (1.19) | 21.4 (1.4)
  6 weeks | 22.13 (1.15) | 21.36 (1.2)
  12 weeks | 21.42 (1.28) | 22.93 (1.3)

14. Primary Outcome: Sexual Function as Assessed by the Watts Sexual Function Questionnaire (WSFQ), Erectile Function
Description: The domain of erectile function/orgasm consists of 7 items. A five-point Likert-type scale ranging from "always" to "never" is used to generate a score, ranging from 7-35. Higher scores indicate increased erectile function/achievement of orgasm.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 26.83 (1.35) | 26 (1.24)
  6 weeks | 26.29 (1.14) | 25.92 (1.44)
  12 weeks | 25.36 (1.65) | 27.46 (1.5)

15. Primary Outcome: Sexual Function as Assessed by the Watts Sexual Function Questionnaire (WSFQ), Arousal
Description: The domains of arousal (1 item subscale of the WSFQ), is assessed using a five-point Likert-type scale ranging from "always" to "never" to generate the score for arousal. The higher the number (range 1-5), the more the participant is able to experience arousal.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 3.92 (0.33) | 3.79 (0.37)
  6 weeks | 4.36 (0.23) | 4.13 (0.27)
  12 weeks | 3.45 (0.51) | 4.31 (0.31)

16. Primary Outcome: Sexual Function as Assessed by the Watts Sexual Function Questionnaire (WSFQ), Sanctification
Description: The domains of satisfaction (3 items), is assessed using a five-point Likert-type scale ranging from "always" to "never" to generate the score, ranging from 3-15. The higher the number, the higher the level of satisfaction with sexual function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 10.92 (0.77) | 10.69 (0.71)
  6 weeks | 11 (0.71) | 11.92 (0.81)
  12 weeks | 11.75 (0.68) | 12.5 (0.69)

17. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Total Score
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. A score of 0-5 is awarded to each of the 15 questions which refer to the past 4 weeks only. The questions are split into the 4 main domains of male sexual function: erectile function, orgasmic function, sexual desire and intercourse satisfaction. The total score ranges from 6-75 with 6 being minimal erectile function and 75 representing maximal erectile function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 21.33 (5.17) | 11.31 (2.1)
  6 weeks | 17.4 (4.6) | 13.2 (2.24)
  12 weeks | 17.08 (5) | 15 (3.29)

18. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Erectile Function
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials. Erectile function is one domain, making up 6 out of 15 questions. The score ranges from 1-30, with the lowest score representing minimal erectile function.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 7.33 (2.44) | 3.27 (1.07)
  6 weeks | 5.87 (2.35) | 3.67 (1.06)
  12 weeks | 5.85 (2.44) | 4.53 (1.55)

19. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Intercourse Satisfaction
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials, one domain being satisfaction with intercourse. A score of 0-5 is awarded to each of the 3 questions which refer to the past 4 weeks only. The score rangers from 0-15, with a score of 0 indicating that no intercourse was attempted in the last 4 weeks, 1= almost or little to no sanctification, 15= very highly satisfied.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 3.8 (1.35) | 0.67 (0.46)
  6 weeks | 2.33 (1.11) | 1.2 (0.59)
  12 weeks | 2.15 (1.25) | 1.53 (0.74)

20. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Orgasmic Function
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials, one domain being satisfaction with orgasm. A score of 0-5 is awarded to each of the 2 questions which refer to the past 4 weeks only. The score rangers from 1-10, with a score of 0 indicating that no sexual stimulation or intercourse was attempted in the last 4 weeks, 1= almost never or never ejaculated, 10= almost always or always
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 1.73 (0.62) | 0.47 (0.26)
  6 weeks | 1.27 (0.54) | 1.07 (0.5)
  12 weeks | 1.46 (0.87) | 1.13 (0.47)

21. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Sexual Desire
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials, one domain being sexual desire. A score of 0-5 is awarded to each of the 2 questions which refer to the past 4 weeks only. The score rangers from 2-10, with a score of 2 indicating very low or none at all, and 10 representing almost always/very high.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 3.73 (0.6) | 2.8 (0.26)
  6 weeks | 3.47 (0.52) | 3.07 (0.33)
  12 weeks | 3.54 (0.57) | 2.93 (0.34)

22. Primary Outcome: Sexual Function as Assessed by the International Index of Erectile Function (IIEF) Questionnaire, Overall Sexual Satisfaction
Description: IIEF Questionnaire is used for the clinical assessment of erectile dysfunction and treatment outcomes in clinical trials, one domain being sexual satisfaction. A score of 0-5 is awarded to each of the 2 questions which refer to the past 4 weeks only. The score rangers from 2-10, with a score of 2 indicating very dissatisfied and 10 being very satisfied.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 4.73 (0.73) | 3.85 (0.66)
  6 weeks | 4.47 (0.72) | 4.2 (0.63)
  12 weeks | 4.08 (0.61) | 4.64 (0.86)

23. Primary Outcome: Daytime Sleepiness as Assessed by Epworth Sleepiness Scale (ESS)
Description: The ESS is a self-administered questionnaire with 8 questions. Respondents are asked to rate, on a 4-point scale (0-3), their usual chances of dozing off or falling asleep while engaged in eight different activities. Most people engage in those activities at least occasionally, although not necessarily every day. The ESS score (the sum of 8 item scores, 0-3) can range from 0 to 24. The higher the ESS score, the higher that person's average sleep propensity in daily life (ASP), or their 'daytime sleepiness'.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 7.07 (0.928) | 8.2 (1.284)
  6 weeks | 7.2 (0.634) | 7.2 (1.36)
  12 weeks | 7.31 (1.195) | 7.4 (1.05)

24. Primary Outcome: Hot Flashes as Assessed by the Blatt-Kuppermann Index (Hot Flash Component)
Description: Hot flashes were assessed using symptom severity 0= none, slight=1, moderate=2, and severe = 3. Hot flashes have a weighting factor of 4 on the overall Blatt-Kuppermann index, making score ranges 0-12, with 12 being the most severe hot flashes.
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 4.53 (0.729) | 7 (0.941)
  6 weeks | 5 (1.013) | 6.43 (1.212)
  12 weeks | 4.38 (0.903) | 7 (0.845)

25. Primary Outcome: Mental Health as Assessed by the Short Form 36 Questionnaire
Description: The SF-36 has eight scaled scores; the scores are weighted sums of the questions in each section. Scores range from 0 - 100 Lower scores = more disability, higher scores = less disability Sections: Vitality, Physical functioning, Bodily pain, General health perception, Physical role functioning, Emotional role functioning, Social role functioning, Mental health
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 81.23 (4.62) | 69.67 (7.16)
  6 weeks | 77.37 (4.64) | 71.36 (5.62)
  12 weeks | 80.66 (4.87) | 77.18 (4.02)

26. Primary Outcome: Physical Health as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 76.25 (5.59) | 64.25 (6.17)
  6 weeks | 74.73 (4.38) | 65.75 (6.56)
  12 weeks | 72.36 (5.45) | 66.92 (5.63)

27. Primary Outcome: Fatigue as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 64 (5.65) | 50.67 (8.24)
  6 weeks | 63.67 (4.1) | 49.67 (7.28)
  12 weeks | 67.69 (4.62) | 54 (5.88)

28. Primary Outcome: Physical Functioning as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 83.33 (5.53) | 71.67 (9.41)
  6 weeks | 82.14 (4.41) | 71.33 (6.96)
  12 weeks | 84.23 (3.34) | 78.33 (8.07)

29. Primary Outcome: Body Pain as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 78 (5.37) | 66 (6.2)
  6 weeks | 74.33 (5.93) | 73 (7.33)
  12 weeks | 76.35 (5.31) | 74 (6.48)

30. Primary Outcome: General Health Perceptions as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 63.37 (5.24) | 56 (3.94)
  6 weeks | 65.67 (4.57) | 57 (6.15)
  12 weeks | 61.54 (5.2) | 58.67 (4.77)

31. Primary Outcome: Role Limitations Due to Physical Health as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 80 (9.82) | 63.33 (11.67)
  6 weeks | 71.67 (9.41) | 61.67 (11.41)
  12 weeks | 67.31 (12.46) | 56.67 (10.76)

32. Primary Outcome: Role Limitations Due to Emotional Role Functioning as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 82.22 (9.12) | 68.89 (11.02)
  6 weeks | 75.56 (10.01) | 75.56 (8.27)
  12 weeks | 76.92 (10.93) | 80 (7.83)

33. Primary Outcome: Social Functioning Due to Emotional Role Functioning as Assessed by the Short Form 36 Questionnaire
Description: as for outcome 25
Time Frame: baseline, 6 weeks, 12 weeks
Measure: Mean (Standard Deviation); unit: units on a scale
Arm/Group | Placebo | Isoflavone
Number analyzed (Participants) | 16 | 17
units on a scale
  Baseline | 94.17 (4.2) | 78.33 (9)
  6 weeks | 83.33 (6.06) | 78.33 (8.75)
  12 weeks | 89.42 (3.7) | 88.33 (5.38)

ADVERSE EVENTS:
Arm/Group | Isoflavone | Placebo
All-Cause Mortality (participants affected / at risk) | 0/17 | 0/16
Serious Adverse Events (participants affected / at risk) | 0/17 | 0/16
Other Adverse Events (participants affected / at risk) | 0/17 | 0/16

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: Yes